CLINICAL TRIAL: NCT07054801
Title: Intra-arterial Lidocaine and Methylprednisolone Injection Into the Middle Meningeal Artery For Treatment of Headache Associated With Subarachnoid Hemorrhage
Brief Title: IA Lidocaine and Methylprednisolone for Headache Associated With Subarachnoid Hemorrhage
Acronym: LIMSAH
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daniel Raper, MBBS (Other)
Responsible Party: Sponsor-Investigator, Daniel Raper, MBBS, Assistant Professor, Neurological Surgery, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-40755
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Headaches Associated With Subarachnoid Hemorrhage (SAH)
Keywords: Headache; Subarachnoid hemorrhage; Lidocaine; Methylprednisolone; Intra-arterial; Middle meningeal artery; Digital subtraction angiography
MeSH Terms: conditions — Headache; Subarachnoid Hemorrhage | interventions — Lidocaine; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Cohort (Experimental): Intra-arterial 80 mg lidocaine and 40 mg methylprednisolone
  Interventions: Drug: Lidocaine hydrochloride; Drug: Methylprednisolone sodium succinate

INTERVENTIONS:
Drug: Lidocaine hydrochloride — A total of 20 mg injected in 10 mg doses will be administered over 5 min into the frontal and parietal branches of each MMA, resulting in a cumulative dose of 40 mg per MMA. The injection will be performed bilaterally, yielding a total dose of 80 mg per patient.
  Other Names: Xylocaine-MPF
Drug: Methylprednisolone sodium succinate — A total of 10 mg were injected over 5 min into the frontal and parietal branches of each MMA, resulting in a cumulative dose of 20 mg per MMA, yielding a total dose of 40 mg per patient.
  Other Names: Solu-MEDROL

SUMMARY:
Subarachnoid hemorrhage (SAH) is a type of bleeding around the brain that can cause sudden and severe headaches. These headaches can be debilitating and persist for weeks, significantly impacting a patient's comfort and recovery. Many patients require opioids for pain control, which can lead to side effects such as drowsiness, constipation, and dependency. There is a need for new treatment strategies to help relieve this pain while minimizing side effects.

This clinical study is designed to evaluate whether an injection of two medications (lidocaine and methylprednisolone) directly into the middle meningeal artery (MMA) can help reduce headache severity in patients who recently experienced a SAH. The medications will be given through a minimally invasive procedure performed during a routine angiogram, a type of imaging test already commonly used in SAH patients. The main goals of the study are to determine whether this treatment approach is safe, helps to reduce the severity of headaches, and decreases the need for opioid pain medications. Eligible patients will be those recently diagnosed with persistent headache symptoms and SAH who are undergoing routine cerebral angiogram, during which the medications are infused into the MMA. Participants will be monitored for pain levels using the Headache Impact Test (HIT-6) and for changes in their functional recovery using standard neurologic scales. The results of this study may provide early evidence to support new treatment options for patients suffering from difficult-to-control headaches after a SAH.

DETAILED DESCRIPTION:
This is a single-center, prospective, single-arm, open-label clinical trial evaluating the safety and efficacy of intra-arterial administration of lidocaine and methylprednisolone sodium succinate via the MMA for the treatment of moderate or severe headaches associated with SAH. Eligible participants will include adult patients diagnosed with SAH who are undergoing diagnostic or therapeutic digital subtraction angiography (DSA). During the DSA procedure, following routine angiographic imaging, a microcatheter will be placed in the MMA, and a low dose of lidocaine and methylprednisolone will be slowly infused under fluoroscopic guidance.

The primary outcome will assess the change in headache severity using the HIT-6 score at baseline (pre-intervention), discharge, and at 1, 6, and 12 weeks postoperatively. Secondary outcomes will include reduction in opioid use, neurological outcome measured by the modified Rankin Scale at discharge and follow-up, and the incidence of any adverse events related to the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥18 years with confirmed SAH via computed tomography or magnetic resonance imaging
2. Undergoing DSA as part of routine diagnostic or therapeutic care
3. Experiencing headaches with baseline severity assessable using Headache Impact Test (HIT-6) questionnaire and 11-point Numeric Rating Scale (NRS)
4. Conscious patients who can understand and sign informed consent form
5. Hemodynamically stable and suitable for intra-arterial procedures

5) Willingness to comply with study procedures and follow-ups

Exclusion Criteria:

1. Known allergy or hypersensitivity to lidocaine or amide-type anesthetics
2. Known allergy or hypersensitivity to Intralipid® (intravenous fat emulsion) or any of its components, including egg phospholipids or soy-based products
3. Known allergy or hypersensitivity to methylprednisolone, corticosteroids, any component of the Solu-Medrol® formulation
4. Diagnostic abnormalities at baseline, including ECG abnormalities (e.g., prolonged PR/QTc intervals, heart block, arrhythmias)
5. Cardiac conditions including history of heart block, Stokes-Adams syndrome, Wolff-Parkinson-White syndrome, or use of antiarrhythmics
6. Steroid-induced psychiatric history; uncontrolled seizures; uncontrolled diabetes; glaucoma/ocular hypertension; current/recent high-dose systemic steroids.
7. Previous IA lidocaine or methylprednisolone (or similar) therapy prior to enrollment
8. Alternative headache etiology (e.g., migraines, tension-type headache)
9. Unable to report pain reliably due to severe cognitive or communication deficits
10. Severe hemodynamic instability precluding safe DSA participation
11. Contraindications to IA catheterization or DSA (e.g., severe peripheral vascular disease, contrast allergies)
12. Severe renal impairment (eGFR <30 mL/min/1.73 m²)
13. Severe hepatic impairment (e.g., Child-Pugh Class C)
14. Active systemic infections
15. Severe comorbid conditions with life expectancy <30 days
16. Participants who are pregnant or breastfeeding
17. Conditions or concomitant medications listed in the USPI for study drugs that would compromise safety or data quality
18. Current participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Headache Severity | From baseline to 12-week follow-up
  Headache Impact Test-6 (HIT-6) score from baseline (pre-intervention) to 12 weeks postoperatively. Scores range from 36 (no impact) to 78 (severe impact), with higher scores indicating a greater negative impact.

SECONDARY OUTCOMES:
Headache intensity | From baseline to 12-week follow-up
  11-point Numeric Rating Scale (NRS) score from baseline (pre-intervention) to 12 weeks postoperatively. Scores range from 0 (no pain) to 10 (worst possible pain), with higher scores indicating a greater negative impact.
Opioid Use | From admission to 12-week follow-up
  Total opioid use will be recorded during hospital stay and follow-up.
Functional Outcome | From discharge to 12-week follow-up
  Functional status will be assessed using the modified Rankin Scale at discharge and follow-up. Scores range from 0 (no symptoms) to 6 (death), with lower scores indicating better outcomes.
Adverse Events Related to Intra-Arterial Injection | From discharge to 12-week follow-up
  All procedural and post-procedural complications will be monitored, including symptoms of lidocaine toxicity, new neurological deficits, worsening headache, hemodynamic instability, or allergic reactions. Events will be categorized by severity and attribution to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Raper, MBBS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No